CLINICAL TRIAL: NCT01451866
Title: Comparison of a Classic Leg-press Training Compared to a Complex Training on a Dynamic Leg-press With Visual Feed-back. Pilot-study
Brief Title: Comparison Between Classic Leg-press Training and Complex Leg-press Training on a Dynamic Leg-press
Acronym: dlp
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Principal Investigator, Roger Hilfiker, Director of Bachelor Thesis, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BA09_DLP
Record Dates: First submitted 2011-09-26; First posted 2011-10-14 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: resistance training; Healthy People Programs
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- classic leg-press training (Active Comparator): Classic resistance training on the dynamic leg press. 6 x 8 repetitions at 60% 1 RM
  Interventions: Other: resistance training
- Complex leg-press training (Experimental): Complex leg-press training with visual feed-back on a dynamic leg-press.
  Interventions: Other: complex resistance training

INTERVENTIONS:
Other: resistance training — hypertrophic resistance training
  Arms: classic leg-press training
Other: complex resistance training — complex resistance training with speed, excentric and power-endurance elements
  Arms: Complex leg-press training

SUMMARY:
A complex training on a dynamic leg-press with visual feed-back will improve coordinative capacity, power, sensorimotor and cognitive aspects more than a classic training on the same leg-press but without visual feed-back.

DETAILED DESCRIPTION:
The project evaluates two different resistance training programs on a leg press. One group will perform a standard resistance training with the aim of muscle hypertrophia, the other group will perform a complex resistance training combining rate of force development training, power training, speed endurance as well as sensorimotor aspects (i.e. following visual feedback to reproduce given forces or joint angles).

Hypotheses: Participants in the complex training group will change the relation between counter movement jump and squat jump, i.e. they will more improve in the counter movement jump because of improved sensorimotor capacity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (>18yrs) participants
* Able to do resistance training

Exclusion Criteria:

* Recent injuries preventing resistance training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
coordination | 5 weeks
  coordination, i.e. sensorimotor capacity measured with (a) the difference between counter-movement jump and squat jump and (b) with a test for dynamic joint-position sense on the dynamic leg press

SECONDARY OUTCOMES:
Power | 5 weeks
  power measured on the dynamic leg press and with the squat jumps
Balance | 5 weeks
  Balance measured with the Star Excursion Balance Test
Power - Endurance | 5 weeks
  Repeated power production during a repeated chair rise test where participants rise from a chair during one minute with two second rest between rises.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Hilfiker, MPTSc., Study Chair — HES-SO Valais
Locations (1):
- Swiss Olympic Medical Center Leukerbad, Leukerbad, Valais, Switzerland